CLINICAL TRIAL: NCT01980940
Title: A Study to Assess the Single Dose Pharmacokinetics of Two and Proof of Efficacy of One New Etoricoxib Gel Formulation in Osteoarthritis Patients
Brief Title: The Single Dose Pharmacokinetics of Two and Proof of Efficacy of One New Etoricoxib Gel Formulation in Participants With Osteoarthritis (MK-0663-168)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0663-168
Record Dates: First submitted 2013-11-05; First posted 2013-11-11 (Estimated); Results first posted 2015-12-11 (Estimated); Last update posted 2024-06-27 (Actual); Status verified 2022-02

CONDITIONS: Osteoarthritis Pain
MeSH Terms: interventions — Etoricoxib; Dimethyl Sulfoxide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Pt 1: ETOR 75 DMSO/ETOR 150 PG/ETOR 75 PG/ETOR 150 DMSO (Experimental): Single-dose etoricoxib 75 mg (1.97 mL) 4% DMSO gel, followed by single-dose etoricoxib 150 mg (4.30 mL) 4% PG gel, followed by single-dose etoricoxib 75 mg (2.15 mL) 4% PG gel, followed by single-dose etoricoxib 150 mg (3.94 mL) 4% DMSO gel. All treatments were applied topically.
  Interventions: Drug: Etoricoxib 75 mg 4% DMSO Gel; Drug: Etoricoxib 75 mg 4% PG Gel; Drug: Etoricoxib 150 mg 4% DMSO Gel; Drug: Etoricoxib 150 mg 4% PG Gel
- Pt 1: ETOR 75 PG/ETOR 75 DMSO/ETOR 150 DMSO/ETOR 150 PG (Experimental): Single-dose etoricoxib 75 mg (2.15 mL) 4% PG gel, followed by single-dose etoricoxib 75 mg (1.97 mL) 4% DMSO gel, followed by single-dose etoricoxib 150 mg (3.94 mL) 4% DMSO gel, followed by single-dose etoricoxib 150 mg (4.30 mL) 4% PG gel. All treatments were applied topically.
  Interventions: Drug: Etoricoxib 75 mg 4% DMSO Gel; Drug: Etoricoxib 75 mg 4% PG Gel; Drug: Etoricoxib 150 mg 4% DMSO Gel; Drug: Etoricoxib 150 mg 4% PG Gel
- Pt 1: ETOR 150 DMSO/ETOR 75 PG/ETOR 150 PG/ETOR 75 DMSO (Experimental): Single-dose etoricoxib 150 mg (3.94 mL) 4% DMSO gel, followed by single-dose etoricoxib 75 mg (2.15 mL) 4% PG gel, followed by single-dose etoricoxib 150 mg (4.30 mL) 4% PG gel, followed by single-dose etoricoxib 75 mg (1.97 mL) 4% DMSO gel. All treatments were applied topically.
  Interventions: Drug: Etoricoxib 75 mg 4% DMSO Gel; Drug: Etoricoxib 75 mg 4% PG Gel; Drug: Etoricoxib 150 mg 4% DMSO Gel; Drug: Etoricoxib 150 mg 4% PG Gel
- Pt 1: ETOR 150 PG/ETOR 150 DMSO/ETOR 75 PG/ETOR 75 DMSO (Experimental): Single-dose etoricoxib 150 mg (4.30 mL) 4% PG gel, followed by single-dose etoricoxib 150 mg (3.94 mL) 4% DMSO gel, followed by single-dose etoricoxib 75 mg (1.97 mL) 4% DMSO gel, followed by single-dose etoricoxib 75 mg (2.15 mL) 4% PG gel. All treatments were applied topically.
  Interventions: Drug: Etoricoxib 75 mg 4% DMSO Gel; Drug: Etoricoxib 75 mg 4% PG Gel; Drug: Etoricoxib 150 mg 4% DMSO Gel; Drug: Etoricoxib 150 mg 4% PG Gel
- Pt 1: ETOR OD/ ETOR 150 DMSO/ ETOR 75 DMSO/ ETOR 75 PG (Experimental): Single-dose etoricoxib 163 mg (4.30 mL) 4% DMSO gel (DMSO formulation administered in error/overdose [OD]), followed by single-dose etoricoxib 150 mg (3.94 mL) 4% DMSO gel, followed by single-dose etoricoxib 75 mg (1.97 mL) 4% DMSO gel, followed by single-dose etoricoxib 75 mg (2.15 mL) 4% PG gel. All treatments were applied topically.
  Interventions: Drug: Etoricoxib 75 mg 4% DMSO Gel; Drug: Etoricoxib 75 mg 4% PG Gel; Drug: Etoricoxib 150 mg 4% DMSO Gel; Drug: Etoricoxib 163 mg 4% DMSO gel
- Pt 1: Placebo (Deviation) (Other): Participants randomized to a treatment sequence in Part 1 who received single dose placebo gel (1.97 or 3.94 mL) applied topically in error instead of active study drug and dropped out after the first treatment period in the sequence. Included in the safety assessments only.
  Interventions: Drug: Placebo
- Pt 2: ETOR 50 DMSO (Experimental): Etoricoxib 50 mg (1.31 mL, 4% DMSO gel) applied topically twice daily to the affected knee for a period of 2 weeks.
  Interventions: Drug: Etoricoxib 50 mg 4% DMSO
- Pt 2: Placebo (Placebo Comparator): Matching placebo to etoricoxib 50 mg 1.31 mL 4% DMSO gel applied topically twice daily to the affected knee for a period of 2 weeks.
  Interventions: Drug: Matching Placebo to Etoricoxib 50 mg 4% DMSO Gel

INTERVENTIONS:
Drug: Etoricoxib 75 mg 4% DMSO Gel — Etoricoxib 75 mg 4% DMSO gel applied topically.
  Arms: Pt 1: ETOR 150 DMSO/ETOR 75 PG/ETOR 150 PG/ETOR 75 DMSO; Pt 1: ETOR 150 PG/ETOR 150 DMSO/ETOR 75 PG/ETOR 75 DMSO; Pt 1: ETOR 75 DMSO/ETOR 150 PG/ETOR 75 PG/ETOR 150 DMSO; Pt 1: ETOR 75 PG/ETOR 75 DMSO/ETOR 150 DMSO/ETOR 150 PG; Pt 1: ETOR OD/ ETOR 150 DMSO/ ETOR 75 DMSO/ ETOR 75 PG
Drug: Etoricoxib 75 mg 4% PG Gel — Etoricoxib 75 4% PG gel applied topically.
  Arms: Pt 1: ETOR 150 DMSO/ETOR 75 PG/ETOR 150 PG/ETOR 75 DMSO; Pt 1: ETOR 150 PG/ETOR 150 DMSO/ETOR 75 PG/ETOR 75 DMSO; Pt 1: ETOR 75 DMSO/ETOR 150 PG/ETOR 75 PG/ETOR 150 DMSO; Pt 1: ETOR 75 PG/ETOR 75 DMSO/ETOR 150 DMSO/ETOR 150 PG; Pt 1: ETOR OD/ ETOR 150 DMSO/ ETOR 75 DMSO/ ETOR 75 PG
Drug: Etoricoxib 150 mg 4% DMSO Gel — Etoricoxib 150 mg 4% DMSO gel applied topically.
  Arms: Pt 1: ETOR 150 DMSO/ETOR 75 PG/ETOR 150 PG/ETOR 75 DMSO; Pt 1: ETOR 150 PG/ETOR 150 DMSO/ETOR 75 PG/ETOR 75 DMSO; Pt 1: ETOR 75 DMSO/ETOR 150 PG/ETOR 75 PG/ETOR 150 DMSO; Pt 1: ETOR 75 PG/ETOR 75 DMSO/ETOR 150 DMSO/ETOR 150 PG; Pt 1: ETOR OD/ ETOR 150 DMSO/ ETOR 75 DMSO/ ETOR 75 PG
Drug: Etoricoxib 150 mg 4% PG Gel — Etoricoxib 150 mg 4% PG gel applied topically.
  Arms: Pt 1: ETOR 150 DMSO/ETOR 75 PG/ETOR 150 PG/ETOR 75 DMSO; Pt 1: ETOR 150 PG/ETOR 150 DMSO/ETOR 75 PG/ETOR 75 DMSO; Pt 1: ETOR 75 DMSO/ETOR 150 PG/ETOR 75 PG/ETOR 150 DMSO; Pt 1: ETOR 75 PG/ETOR 75 DMSO/ETOR 150 DMSO/ETOR 150 PG
Drug: Etoricoxib 163 mg 4% DMSO gel — Etoricoxib 163 mg 4% DMSO gel applied topically
  Arms: Pt 1: ETOR OD/ ETOR 150 DMSO/ ETOR 75 DMSO/ ETOR 75 PG
Drug: Placebo — Placebo gel applied topically.
  Arms: Pt 1: Placebo (Deviation)
Drug: Etoricoxib 50 mg 4% DMSO — Etoricoxib 50 mg 4% DMSO gel applied topically.
  Arms: Pt 2: ETOR 50 DMSO
Drug: Matching Placebo to Etoricoxib 50 mg 4% DMSO Gel — Matching Placebo to Etoricoxib 50 mg 4% DMSO gel applied topically.
  Arms: Pt 2: Placebo

SUMMARY:
Study Part 1 is designed to assess the plasma pharmacokinetics of etoricoxib (ETOR) 4% dimethyl sulfoxide (DMSO) and propylene glycol (PG) formulations, each at 2 different doses, upon single-dose topical administration on the knee of osteoarthritis participants. Study Part 2 is designed to evaluate the efficacy of topical etoricoxib vs. placebo in the treatment of osteoarthritis of the knee. The primary hypothesis is that topical etoricoxib will be more effective than placebo in the treatment of osteoarthritis of the knee over 2 weeks of treatment as assessed by time-weighted average change from baseline on the Western Ontario and McMaster Universities Arthritis Index (WOMAC) Visual Analogue (VA) 3.0 pain subscale.

DETAILED DESCRIPTION:
Part I of the study will consist of a single-dose, open-label, randomized, four-way cross over study with topical administration of etoricoxib gel on the knee of osteoarthritis participants. The washout between successive dose administrations will be at least one week. Part 2 of the study will consist of double-blind, randomized, placebo-controlled, parallel groups, multiple dose, twice daily topical administration of etoricoxib or placebo gel on the knee of osteoarthritis participants for a period of two weeks.

ELIGIBILITY:
Inclusion Criteria

* Has diagnosis of osteoarthritis of the knee (tibio-femoral joint) for >6 months based on clinical and radiographic criteria;
* Has a diagnosis of American Rheumatology Association (ARA) functional Class I, II, or III;
* The knee designated as the "study joint" must be the participant's primary source of pain/disability in the lower extremity. If both knees are affected, the most painful joint will be selected for evaluation for inclusion and clinical response;
* Female participants of childbearing potential must demonstrate a serum beta human chorionic gonadotropin (β-hCG) level consistent with a non-gravid state at the screening visit and urine β-hCG at Day -1 prior to first dosing and agree to use adequate oral or barrier contraception or abstain from sexual contact at least 7 days prior to treatment and continuing through the treatment period or a discontinuation visit;
* Willing to limit alcohol intake (beer 8 ounces, wine 4 ounces, liquor 1 ounce) to no more than 14 drinks a week (no more than 2 in a day) and to avoid unaccustomed strenuous physical activity (e.g., unaccustomed weight lifting, initiation of physical therapy) for the duration of the study;
* Judged to be in general good health with the exception of osteoarthritis based on medical history, physical examination, and routine laboratory tests.
* For Part 2, if the participant is a regular user of non-steroidal anti-inflammatory drugs (NSAIDs) including coxibs he/she must report a history of positive therapeutic benefit in osteoarthritis of the knee with NSAID/coxibs in the past;
* For Part 2, participants must be taking a single NSAID on a regular basis and at a prescription strength for at least 30 days prior to study screening ("regular basis" is defined as at least 25 of the previous 30 days) for treatment of symptoms of osteoarthritis.

Exclusion Criteria:

* Has a concurrent medical/arthritic disease;
* History of acute ligamentous or meniscal injury of the study joint within the previous 2 years or arthroscopy of the affected knee within 6 months prior to study entry;
* Is a candidate for imminent joint replacement;
* Has clinical or laboratory evidence of significant renal, gastrointestinal, pulmonary, hepatic, endocrine, neurological (apart from migraine), or other systemic disease that in the opinion of the investigator contraindicates the use of etoricoxib;
* Has congestive heart failure with symptoms that occur at rest or minimal activity;
* Has unstable angina that occurs at rest or with minimal activity;
* Has uncontrolled hypertension (sitting diastolic blood pressure >95 mm Hg, or sitting systolic blood pressure >165 mm Hg);
* Has a history of stroke or transient ischemic attack (TIA) within the previous 6 months;
* Has a history of hepatitis/hepatic disease that has been active within the previous 2 years;
* Has a history of neoplastic disease;
* Is currently a user (including "recreational use") of any illicit drugs, or has a history of drug or alcohol abuse within the past 5 years;
* Is allergic of has hypersensitivity to aspirin, ibuprofen, rofecoxib, celecoxib, valdecoxib, other NSAIDs, acetaminophen, or sulfa drugs;
* Has used intravenous, intramuscular, or oral corticosteroids within 1 month of study entry;
* Has used glucosamine and/or chondroitin sulfate for <6 months prior to study start;
* Has used intra-articular steroids, HYALGAN™ (sodium hyaluronate, Sanofi Pharmaceuticals), or SYNVISC™ (hylan G-F 20, Wyeth-Ayerst Pharmaceuticals) to the study joint within 3 months of entry into the study or intra-articular steroids, HYALGAN™, or SYNVISC™ to any other joint within 1 month of study entry;
* Has used topical, oral or systemic analgesic medications within 2 weeks of study entry and for the duration of the study;
* Requires treatment with warfarin, heparin, high-dose aspirin (>325 mg), or digoxin;
* Has used Arcoxia® within 2 weeks of study entry.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-12-23 (Actual); Primary Completion 2014-11-26 (Actual); Study Completion 2014-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were screened for inclusion in the study over 4 weeks prior to first treatment. Two additional participants were screened for Study Part 1 but not randomized or treated due to screen failure.
Groups:
- Pt 1: ETOR OD/ ETOR 150 DMSO/ ETOR 75 DMSO/ ETOR 75 PG: Single-dose etoricoxib 163 mg (4.30 mL) 4% DMSO gel (DMSO formulation administered in error/overdose), followed by single-dose etoricoxib 150 mg (3.94 mL) 4% DMSO gel, followed by single-dose etoricoxib 75 mg (1.97 mL) 4% DMSO gel, followed by single-dose etoricoxib 75 mg (2.15 mL) 4% PG gel. All treatments were applied topically.
Period: Overall Study
Arm/Group | Pt 1: ETOR 75 DMSO/ETOR 150 PG/ETOR 75 PG/ETOR 150 DMSO | Pt 1: ETOR 75 PG/ETOR 75 DMSO/ETOR 150 DMSO/ETOR 150 PG | Pt 1: ETOR 150 DMSO/ETOR 75 PG/ETOR 150 PG/ETOR 75 DMSO | Pt 1: ETOR 150 PG/ETOR 150 DMSO/ETOR 75 PG/ETOR 75 DMSO | Pt 1: ETOR OD/ ETOR 150 DMSO/ ETOR 75 DMSO/ ETOR 75 PG | Pt 1: Placebo (Deviation) | Pt 2: ETOR 50 DMSO | Pt 2: Placebo
Started | 5 | 5 | 5 | 3 | 2 | 2 | 24 | 24
Treated | 5 | 5 | 5 | 3 | 2 | 2 | 24 | 24
Completed | 5 | 5 | 5 | 3 | 2 | 0 | 24 | 24
Not Completed | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pt 1: ETOR 75 DMSO/ETOR 150 PG/ETOR 75 PG/ETOR 150 DMSO | Pt 1: ETOR 75 PG/ETOR 75 DMSO/ETOR 150 DMSO/ETOR 150 PG | Pt 1: ETOR 150 DMSO/ETOR 75 PG/ETOR 150 PG/ETOR 75 DMSO | Pt 1: ETOR 150 PG/ETOR 150 DMSO/ETOR 75 PG/ETOR 75 DMSO | Pt 1: ETOR OD/ ETOR 150 DMSO/ ETOR 75 DMSO/ ETOR 75 PG | Pt 1: Placebo (Deviation) | Pt 2: ETOR 50 DMSO | Pt 2: Placebo | Total
Number analyzed (Participants) | 5 | 5 | 5 | 3 | 2 | 2 | 24 | 24 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (6.6) | 61.0 (12.3) | 63.6 (10.6) | 62.0 (10.0) | 55.0 (8.5) | 60.5 (4.9) | 61.5 (8.2) | 61.2 (6.7) | 61.3 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 4 | 3 | 1 | 0 | 18 | 15 | 48
  Male | 1 | 2 | 1 | 0 | 1 | 2 | 6 | 9 | 22

OUTCOME MEASURES:

1. Primary Outcome: Study Part 1: Maximum Concentration (Cmax) of ETOR After Single Dosing
Description: Cmax determined for the period up to 72 hours post-single application. Descriptive statistics are expressed as the geometric least squares mean (GLSM). Cmax with value 0 included in calculation of GLSMs with a value of 0.5*LLOQ (=0.5 h*ng/ml).
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 7, 9, 12, 16, 24, 36, 48, and 72 hours post-application
Population: PK analysis set defined as all participants treated with etoricoxib with sufficient PK data for reliable estimation of the PK parameter of interest (Cmax) without any protocol violation that interferes with PK data interpretation
Measure: Least Squares Mean (90% Confidence Interval); unit: mg
Groups:
- ETOR 75 DMSO: Single-dose etoricoxib 75 mg (1.97 mL) 4% DMSO gel applied topically.
- ETOR 75 PG: Single-dose etoricoxib 75 mg (2.15 mL) 4% PG gel applied topically.
- ETOR 150 DMSO: Single-dose etoricoxib 150 mg (3.94 mL) 4% DMSO gel applied topically.
- ETOR 150 PG: Single-dose etoricoxib 150 mg (4.30 mL) 4% PG gel applied topically.
- ETOR OD: Single-dose etoricoxib 163 mg (4.30 mL) 4% DMSO gel applied topically (DMSO formulation administered in overdose/error).
- Placebo (Pt 1) (Deviation): Single dose placebo (1.97 mL or 3.94 mL) gel applied topically (placebo gel administered in error instead of active study drug formulation).
Arm/Group | ETOR 75 DMSO | ETOR 75 PG | ETOR 150 DMSO | ETOR 150 PG | ETOR OD | Placebo (Pt 1) (Deviation)
Number analyzed (Participants) | 20 | 20 | 20 | 18 | 0 | 0
mg | 12.39 (8.24) [9.95 to 15.43] | 2.43 (2.14) [1.83 to 3.24] | 27.30 (15.30) [22.76 to 32.75] | 3.74 (3.79) [3.00 to 4.66] |  |
Statistical Analysis 1: Comparison: ETOR 75 DMSO vs ETOR 75 PG; The geometric least squares mean ratio (GLSMR) and 90% confidence interval was calculated for Cmax after log transformation for the formulation comparison (ETOR 75 DMSO/ETOR 75 PG) using a linear mixed effect model with fixed effects terms for treatment and period and random effect for participants. Cmax with value 0 included in calculation of GLSMs with a value of 0.5*LLOQ (=0.5 h*ng/ml); Test type: Superiority or Other; ANOVA; Treatment ratio = 5.09, 90% CI 2-sided [4.03 to 6.42]
Statistical Analysis 2: Comparison: ETOR 150 DMSO vs ETOR 150 PG; The GLSMR and 90% confidence interval was calculated for Cmax after log transformation for the formulation comparison (ETOR 150 DMSO/ETOR 150 PG) using a linear mixed effect model with fixed effects terms for treatment and period and random effect for participants. Cmax with value 0 included in calculation of GLSMs with a value of 0.5*LLOQ (=0.5 h*ng/ml); Test type: Superiority or Other; ANOVA; Treatment ratio = 7.30, 90% CI 2-sided [6.05 to 8.81]
Statistical Analysis 3: Comparison: ETOR 75 DMSO vs ETOR 150 DMSO; The GLSMR and 90% confidence interval was calculated for Cmax after log transformation for the dose comparison (ETOR 75 DMSO/ETOR 150 DMSO) using a linear mixed effect model with fixed effects terms for treatment and period and random effect for participants. Cmax with value 0 included in calculation of GLSMs with a value of 0.5*LLOQ (=0.5 h*ng/ml); Test type: Superiority or Other; ANOVA; Treatment ratio = 0.45, 90% CI 2-sided [0.38 to 0.55]
Statistical Analysis 4: Comparison: ETOR 75 PG vs ETOR 150 PG; The GLSMR and 90% confidence interval was calculated for Cmax after log transformation for the dose comparison (ETOR 75 PG/ETOR 150 PG) using a linear mixed effect model with fixed effects terms for treatment and period and random effect for participants. Cmax with value 0 included in calculation of GLSMs with a value of 0.5*LLOQ (=0.5 h*ng/ml); Test type: Superiority or Other; ANOVA; Treatment ratio = 0.65, 90% CI 2-sided [0.51 to 0.83]

2. Primary Outcome: Study Part 1: Time to Maximum Concentration (Tmax) of ETOR After Single Dosing
Description: Tmax determined for the period up to 72 hours post-single application.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 7, 9, 12, 16, 24, 36, 48, and 72 hours post-application
Population: PK analysis set defined as all participants treated with etoricoxib with sufficient PK data for reliable estimation of the PK parameter of interest (Tmax) without any protocol violation that interferes with PK data interpretation
Measure: Median (Full Range); unit: hour
Arm/Group | ETOR 75 DMSO | ETOR 75 PG | ETOR 150 DMSO | ETOR 150 PG | ETOR OD | Placebo (Pt 1) (Deviation)
Number analyzed (Participants) | 20 | 18 | 20 | 18 | 2 | 0
hour | 30.0 [23.5 to 72.0] | 48.0 [1.0 to 72.0] | 24.0 [2.0 to 72.0] | 48 [24.0 to 72.0] | 36.0 [24.0 to 48.0] |

3. Primary Outcome: Study Part 1: Area Under the Concentration-time Curve of ETOR From Time 0 to Last (AUC0-last) After Single Dosing
Description: Area under the observed concentration-time curve from time zero to the last quantifiable time point determined for the period up to 72 hours post-single application. The area was calculated according to the linear up/log down trapezoidal rule. AUC0-last is an estimate of total plasma exposure. Descriptive statistics are expressed as the GLSM. AUC with value 0 included in calculation of GLSMs with a value of 0.5*LLOQ (=0.5 h*ng/ml).
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 7, 9, 12, 16, 24, 36, 48, and 72 hours post-application
Population: PK analysis set defined as all participants treated with etoricoxib with sufficient PK data for reliable estimation of the PK parameter of interest (AUC0-last) without any protocol violation that interferes with PK data interpretation
Measure: Least Squares Mean (90% Confidence Interval); unit: mg
Arm/Group | ETOR 75 DMSO | ETOR 75 PG | ETOR 150 DMSO | ETOR 150 PG | ETOR OD | Placebo (Pt 1) (Deviation)
Number analyzed (Participants) | 20 | 20 | 20 | 18 | 0 | 0
mg | 611.3 (400.97) [493.9 to 756.6] | 65.6 (112.83) [30.7 to 140.0] | 1309.7 (686.34) [1086.0 to 1579.5] | 161.3 (172.96) [122.3 to 212.9] |  |
Statistical Analysis 1: Comparison: ETOR 75 DMSO vs ETOR 75 PG; The GLSMR and 90% confidence interval was calculated for AUC0-last after log transformation for the formulation comparison (ETOR 75 DMSO/ETOR 75 PG) using a linear mixed effect model with fixed effects terms for treatment and period and random effect for participants. AUC with value 0 included in calculation of GLSMs with a value of 0.5*LLOQ (=0.5 h*ng/ml); Test type: Superiority or Other; ANOVA; Treatment ratio = 9.32, 90% CI 2-sided [4.77 to 18.18]
Statistical Analysis 2: Comparison: ETOR 150 DMSO vs ETOR 150 PG; The GLSMR and 90% confidence interval was calculated for AUC0-last after log transformation for the formulation comparison (ETOR 150 DMSO/ETOR 150 PG) using a linear mixed effect model with fixed effects terms for treatment and period and random effect for participants. AUC with value 0 included in calculation of GLSMs with a value of 0.5*LLOQ (=0.5 h*ng/ml); Test type: Superiority or Other; ANOVA; Treatment ratio = 8.12, 90% CI 2-sided [6.39 to 10.32]
Statistical Analysis 3: Comparison: ETOR 75 DMSO vs ETOR 150 DMSO; The GLSMR and 90% confidence interval was calculated for AUC0-last after log transformation for the dose comparison (ETOR 75 DMSO/ETOR 150 DMSO) using a linear mixed effect model with fixed effects terms for treatment and period and random effect for participants. AUC with value 0 included in calculation of GLSMs with a value of 0.5*LLOQ (=0.5 h*ng/ml); Test type: Superiority or Other; ANOVA; Treatment ratio = 0.47, 90% CI 2-sided [0.39 to 0.57]
Statistical Analysis 4: Comparison: ETOR 75 PG vs ETOR 150 PG; The GLSMR and 90% confidence interval was calculated for AUC0-last after log transformation for the dose comparison (ETOR 75 PG/ETOR 150 PG) using a linear mixed effect model with fixed effects terms for treatment and period and random effect for participants. AUC with value 0 included in calculation of GLSMs with a value of 0.5*LLOQ (=0.5 h*ng/ml); Test type: Superiority or Other; ANOVA; Treatment ratio = 0.41, 90% CI 2-sided [0.21 to 0.79]

4. Primary Outcome: Study Part 2: Change From Baseline in Mean Participant Score on the Western Ontario and McMaster Universities Arthritis Index (WOMAC) Visual Analog (VA) 3.1 Pain Scale
Description: The WOMAC VA 3.1 Pain subscale is a self-administered questionnaire assessing lower extremity pain due to osteoarthritis that was completed by participants 2 to 3 hours post morning dose. The WOMAC Pain Subscale had five questions with answers to each item assessed on a 100 mm VA scale (0 = no pain; 100 = extreme pain). The score for each item was summed and the overall score ranged from 0 to 500 (increasing severity). The time weighted average up to day x was calculated as the sum of rectangles under the curve for successive intervals prior to day x as defined by timepoints at which assessments were made. The time weighted change from baseline was calculated. A negative mean change from baseline indicates improvement in pain.
Time Frame: Baseline (Day -1), Day 2, Day 4, Day 7, Day 11, Day 14
Population: Full analysis set (FAS) defined as all treated participants (etoricoxib or placebo) without major entry criteria violation and with at least one valid post-baseline primary efficacy assessment
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- ETOR 50 DMSO: Etoricoxib 50 mg (1.31 mL, 4% DMSO gel) applied topically twice daily to the affected knee for a period of 2 weeks.
- Placebo (Pt 2): Matching placebo to etoricoxib 50 mg 1.31 mL 4% DMSO gel applied topically twice daily to the affected knee for a period of 2 weeks.
Arm/Group | ETOR 50 DMSO | Placebo (Pt 2)
Number analyzed (Participants) | 24 | 24
Units on a scale
  BL to Day 2 | -24.21 (76.88) | -37.21 (101.77)
  BL to Day 4 | -34.29 (69.15) | -43.92 (94.81)
  BL to Day 7 | -45.81 (67.92) | -54.11 (94.11)
  BL to Day 11 | -59.42 (71.12) | -63.60 (90.99)
  BL to Day 14 | -69.60 (75.81) | -72.60 (91.35)
Statistical Analysis 1: Comparison: ETOR 50 DMSO vs Placebo (Pt 2); Treatment difference in mean time-weighted average change from baseline to Day 2 in the WOMAC VA 3.1 pain subscale score (ETOR 50 DMSO - Placebo [Pt 2]) was evaluated using a constrained longitudinal data analysis model that included baseline measurements and time-weighted average at Day 2 in the response variable. The model included terms of visit, visit-by-treatment, and treatment; Test type: Superiority or Other; p = 0.2113, constrained longitudinal data analysis; Mean Difference (Final Values) = -27.3, 90% CI 2-sided [-63.6 to 8.9], Standard Error of Mean 21.57
Statistical Analysis 2: Comparison: ETOR 50 DMSO vs Placebo (Pt 2); Treatment difference in mean time-weighted average change from baseline to Day 4 in the WOMAC VA 3.1 pain subscale score (ETOR 50 DMSO - Placebo [Pt 2]) was evaluated using a constrained longitudinal data analysis model that included baseline measurements and time-weighted average at Day 4 in the response variable. The model included terms of visit, visit-by-treatment, and treatment; Test type: Superiority or Other; p = 0.2548, constrained longitudinal data analysis; Mean Difference (Final Values) = -22.7, 90% CI 2-sided [-55.7 to 10.3], Standard Error of Mean 19.66
Statistical Analysis 3: Comparison: ETOR 50 DMSO vs Placebo (Pt 2); Treatment difference in mean time-weighted average change from baseline to Day 7 in the WOMAC VA 3.1 pain subscale score (ETOR 50 DMSO - Placebo [Pt 2]) was evaluated using a constrained longitudinal data analysis model that included baseline measurements and time-weighted average at Day 7 in the response variable. The model included terms of visit, visit-by-treatment, and treatment; Test type: Superiority or Other; p = 0.2880, constrained longitudinal data analysis; Mean Difference (Final Values) = -21.4, 90% CI 2-sided [-54.9 to 12.0], Standard Error of Mean 19.94
Statistical Analysis 4: Comparison: ETOR 50 DMSO vs Placebo (Pt 2); Treatment difference in mean time-weighted average change from baseline to Day 11 in the WOMAC VA 3.1 pain subscale score (ETOR 50 DMSO - Placebo [Pt 2]) was evaluated using a constrained longitudinal data analysis model that included baseline measurements and time-weighted average at Day 11 in the response variable. The model included terms of visit, visit-by-treatment, and treatment; Test type: Superiority or Other; p = 0.3709, constrained longitudinal data analysis; Median Difference (Final Values) = -17.6, 90% CI 2-sided [-50.4 to 15.1], Standard Error of Mean 19.52
Statistical Analysis 5: Comparison: ETOR 50 DMSO vs Placebo (Pt 2); Treatment difference in mean time-weighted average change from baseline to Day 14 in the WOMAC VA 3.1 pain subscale score (ETOR 50 DMSO - Placebo [Pt 2]) was evaluated using a constrained longitudinal data analysis model that included baseline measurements and time-weighted average at Day 14 in the response variable. The model included terms of visit, visit-by-treatment, and treatment; Test type: Superiority or Other; p = 0.3883, constrained longitudinal data analysis; Mean Difference (Final Values) = -17.3, 90% CI 2-sided [-50.5 to 16.0], Standard Error of Mean 19.81

5. Secondary Outcome: Study Part 2: Change From Baseline in Mean Participant Score on the WOMAC VA 3.1 Stiffness Scale
Description: The WOMAC VA 3.1 Stiffness subscale is a self-administered questionnaire assessing lower extremity stiffness due to osteoarthritis that was completed by participants 2 to 3 hours post morning dose. The WOMAC Stiffness subscale had two questions with answers to each item assessed on a 100 mm VA scale (0 = no stiffness; 100 = extreme stiffness). The score for each item was summed and the overall score ranged from 0 to 200 (increasing severity). The time weighted average up to day x was calculated as the sum of rectangles under the curve for successive intervals prior to day x as defined by timepoints at which assessments were made. The time weighted change from baseline was calculated. A negative mean change from baseline indicates improvement in stiffness.
Time Frame: Baseline (Day -1), Day 2, Day 4, Day 7, Day 11, Day 14
Population: FAS defined as all treated participants (etoricoxib or placebo) without major entry criteria violation and with at least one valid post-baseline primary efficacy assessment
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | ETOR 50 DMSO | Placebo (Pt 2)
Number analyzed (Participants) | 24 | 24
Units on a scale
  BL to Day 2 | -9.17 (37.44) | -16.79 (41.86)
  BL to Day 4 | -14.69 (35.23) | -18.79 (39.29)
  BL to Day 7 | -19.34 (35.75) | -23.08 (37.53)
  BL to Day 11 | -24.44 (34.60) | -26.87 (35.26)
  BL to Day 14 | -29.22 (36.64) | -30.52 (34.33)
Statistical Analysis 1: Comparison: ETOR 50 DMSO vs Placebo (Pt 2); Treatment difference in mean time-weighted average change from baseline to Day 2 in the WOMAC VA 3.1 stiffness subscale score (ETOR 50 DMSO - Placebo [Pt 2]) was evaluated using a constrained longitudinal data analysis model that included baseline measurements and time-weighted average at Day 2 in the response variable. The model included terms of visit, visit-by-treatment, and treatment; Test type: Superiority or Other; p = 0.1383, constrained longitudinal data analysis; Mean Difference (Final Values) = -14.1, 90% CI 2-sided [-29.7 to 1.6], Standard Error of Mean 9.32
Statistical Analysis 2: Comparison: ETOR 50 DMSO vs Placebo (Pt 2); Treatment difference in mean time-weighted average change from baseline to Day 4 in the WOMAC VA 3.1 stiffness subscale score (ETOR 50 DMSO - Placebo [Pt 2]) was evaluated using a constrained longitudinal data analysis model that included baseline measurements and time-weighted average at Day 4 in the response variable. The model included terms of visit, visit-by-treatment, and treatment; Test type: Superiority or Other; p = 0.2380, constrained longitudinal data analysis; Mean Difference (Final Values) = -10.4, 90% CI 2-sided [-24.9 to 4.2], Standard Error of Mean 8.66
Statistical Analysis 3: Comparison: ETOR 50 DMSO vs Placebo (Pt 2); Treatment difference in mean time-weighted average change from baseline to Day 7 in the WOMAC VA 3.1 stiffness subscale score (ETOR 50 DMSO - Placebo [Pt 2]) was evaluated using a constrained longitudinal data analysis model that included baseline measurements and time-weighted average at Day 7 in the response variable. The model included terms of visit, visit-by-treatment, and treatment; Test type: Superiority or Other; p = 0.2691, constrained longitudinal data analysis; Mean Difference (Final Values) = -9.5, 90% CI 2-sided [-23.9 to 4.8], Standard Error of Mean 8.53
Statistical Analysis 4: Comparison: ETOR 50 DMSO vs Placebo (Pt 2); Treatment difference in mean time-weighted average change from baseline to Day 11 in the WOMAC VA 3.1 stiffness subscale score (ETOR 50 DMSO - Placebo [Pt 2]) was evaluated using a constrained longitudinal data analysis model that included baseline measurements and time-weighted average at Day 11 in the response variable. The model included terms of visit, visit-by-treatment, and treatment; Test type: Superiority or Other; p = 0.3246, constrained longitudinal data analysis; Mean Difference (Final Values) = -8.1, 90% CI 2-sided [-21.8 to 5.6], Standard Error of Mean 8.15
Statistical Analysis 5: Comparison: ETOR 50 DMSO vs Placebo (Pt 2); Treatment difference in mean time-weighted average change from baseline to Day 14 in the WOMAC VA 3.1 stiffness subscale score (ETOR 50 DMSO - Placebo [Pt 2]) was evaluated using a constrained longitudinal data analysis model that included baseline measurements and time-weighted average at Day 14 in the response variable. The model included terms of visit, visit-by-treatment, and treatment; Test type: Superiority or Other; p = 0.3881, constrained longitudinal data analysis; Mean Difference (Final Values) = -7.1, 90% CI 2-sided [-20.9 to 6.6], Standard Error of Mean 8.19

6. Secondary Outcome: Study Part 2: Change From Baseline in Mean Participant Score on the WOMAC VA 3.1 Physical Functioning Scale
Description: The WOMAC VA 3.1 Physical Functioning subscale is a self-administered questionnaire assessing lower extremity physical function due to osteoarthritis that was completed by participants 2 to 3 hours post morning dose. The WOMAC Physical Functioning subscale had 17 questions with answers to each item assessed on a 100 mm VA scale (0 = no difficulty; 100 = extreme difficulty). The score for each item was summed and the overall score ranged from 0 to 1700 (increasing severity). The time weighted average up to day x was calculated as the sum of rectangles under the curve for successive intervals prior to day x as defined by timepoints at which assessments were made. The time weighted change from baseline was calculated. A negative mean change from baseline indicates improvement in physical function.
Time Frame: Baseline (Day -1), Day 2, Day 4, Day 7, Day 11, Day 14
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | ETOR 50 DMSO | Placebo (Pt 2)
Number analyzed (Participants) | 24 | 24
Units on a scale
  BL to Day 2 | -117.13 (200.38) | -153.54 (278.66)
  BL to Day 4 | -147.71 (183.07) | -171.35 (272.51)
  BL to Day 7 | -172.94 (186.22) | -199.88 (265.29)
  BL to Day 11 | -214.87 (203.95) | -245.05 (238.05)
  BL to Day 14 | -250.82 (218.72) | -280.29 (233.39)
Statistical Analysis 1: Comparison: ETOR 50 DMSO vs Placebo (Pt 2); Treatment difference in mean time-weighted average change from baseline to Day 2 in the WOMAC VA 3.1 physical function subscale score (ETOR 50 DMSO - Placebo [Pt 2]) was evaluated using a constrained longitudinal data analysis model that included baseline measurements and time-weighted average at Day 2 in the response variable. The model included terms of visit, visit-by-treatment, and treatment; Test type: Superiority or Other; p = 0.4477, constrained longitudinal data analysis; Mean Difference (Final Values) = -52.3, 90% CI 2-sided [-166.8 to 62.3], Standard Error of Mean 68.25
Statistical Analysis 2: Comparison: ETOR 50 DMSO vs Placebo (Pt 2); Treatment difference in mean time-weighted average change from baseline to Day 4 in the WOMAC VA 3.1 physical function subscale score (ETOR 50 DMSO - Placebo [Pt 2]) was evaluated using a constrained longitudinal data analysis model that included baseline measurements and time-weighted average at Day 4 in the response variable. The model included terms of visit, visit-by-treatment, and treatment; Test type: Superiority or Other; p = 0.6084, constrained longitudinal data analysis; Mean Difference (Final Values) = -33.7, 90% CI 2-sided [-143.6 to 76.1], Standard Error of Mean 65.42
Statistical Analysis 3: Comparison: ETOR 50 DMSO vs Placebo (Pt 2); Treatment difference in mean time-weighted average change from baseline to Day 7 in the WOMAC VA 3.1 physical function subscale score (ETOR 50 DMSO - Placebo [Pt 2]) was evaluated using a constrained longitudinal data analysis model that included baseline measurements and time-weighted average at Day 7 in the response variable. The model included terms of visit, visit-by-treatment, and treatment; Test type: Superiority or Other; p = 0.5926, constrained longitudinal data analysis; Mean Difference (Final Values) = -35.2, 90% CI 2-sided [-144.7 to 74.4], Standard Error of Mean 65.25
Statistical Analysis 4: Comparison: ETOR 50 DMSO vs Placebo (Pt 2); Treatment difference in mean time-weighted average change from baseline to Day 11 in the WOMAC VA 3.1 physical function subscale score (ETOR 50 DMSO - Placebo [Pt 2]) was evaluated using a constrained longitudinal data analysis model that included baseline measurements and time-weighted average at Day 11 in the response variable. The model included terms of visit, visit-by-treatment, and treatment; Test type: Superiority or Other; p = 0.5022, constrained longitudinal data analysis; Mean Difference (Final Values) = -42.3, 90% CI 2-sided [-147.2 to 62.6], Standard Error of Mean 62.49
Statistical Analysis 5: Comparison: ETOR 50 DMSO vs Placebo (Pt 2); Treatment difference in mean time-weighted average change from baseline to Day 14 in the WOMAC VA 3.1 physical function subscale score (ETOR 50 DMSO - Placebo [Pt 2]) was evaluated using a constrained longitudinal data analysis model that included baseline measurements and time-weighted average at Day 14 in the response variable. The model included terms of visit, visit-by-treatment, and treatment; Test type: Superiority or Other; p = 0.5125, constrained longitudinal data analysis; Mean Difference (Final Values) = -42.0, 90% CI 2-sided [-149.0 to 64.9], Standard Error of Mean 63.70

7. Secondary Outcome: Study Part 2: Percentage of Participants by Category on Patient Global Assessment of Response to Therapy (PGART)
Description: The PGART is a self-administered questionnaire completed by participants. Participant assessment of response of arthritis to study medication was assessed on a 5-point Likert scale ('very well', 'well', 'fair', 'poor', and 'very poor').
Time Frame: Day 2, Day 4, Day 7, Day 11, Day 14, post-trial (up to Day 28)
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | ETOR 50 DMSO | Placebo (Pt 2)
Number analyzed (Participants) | 24 | 24
Percentage of participants
  Day 2: Very well | 0.0 | 0.0
  Day 2: Well | 20.8 | 33.3
  Day 2: Fair | 25.0 | 25.0
  Day 2: Poor | 37.5 | 33.3
  Day 2: Very poor | 16.7 | 8.3
  Day 4: Very well | 0.0 | 0.0
  Day 4: Well | 20.8 | 33.3
  Day 4: Fair | 45.8 | 37.5
  Day 4: Poor | 29.2 | 25.0
  Day 4: Very poor | 4.2 | 4.2
  Day 7: Very well | 0.0 | 0.0
  Day 7: Well | 25.0 | 37.5
  Day 7: Fair | 50.0 | 37.5
  Day 7: Poor | 25.0 | 25.0
  Day 7: Very poor | 0.0 | 0.0
  Day 11: Very well | 0.0 | 0.0
  Day 11: Well | 37.5 | 50.0
  Day 11: Fair | 45.8 | 37.5
  Day 11: Poor | 16.7 | 12.5
  Day 11: Very poor | 0.0 | 0.0
  Day 14: Very well | 0.0 | 8.3
  Day 14: Well | 54.2 | 50.0
  Day 14: Fair | 41.7 | 33.3
  Day 14: Poor | 4.2 | 8.3
  Day 14: Very poor | 0.0 | 0.0
  Post-trial: Very well | 8.3 | 8.3
  Post-trial: Well | 62.5 | 50.0
  Post-trial: Fair | 29.2 | 29.2
  Post-trial: Poor | 0 | 12.5
  Post-trial: Very poor | 0.0 | 0.0
Statistical Analysis 1: Comparison: ETOR 50 DMSO vs Placebo (Pt 2); Treatment comparison of Day 2 PGART frequencies (ETOR 50 DMSO vs Placebo [Pt 2]) was performed using a two-sided Jonckheere-Terpstra test; Test type: Superiority or Other; p = 0.2632, Jonckheere-Terpstra test
Statistical Analysis 2: Comparison: ETOR 50 DMSO vs Placebo (Pt 2); Treatment comparison of Day 4 PGART frequencies (ETOR 50 DMSO vs Placebo [Pt 2]) was performed using a two-sided Jonckheere-Terpstra test; Test type: Superiority or Other; p = 0.4703, Jonckheere-Terpstra test
Statistical Analysis 3: Comparison: ETOR 50 DMSO vs Placebo (Pt 2); Treatment comparison of Day 7 PGART frequencies (ETOR 50 DMSO vs Placebo [Pt 2]) was performed using a two-sided Jonckheere-Terpstra test; Test type: Superiority or Other; p = 0.5507, Jonckheere-Terpstra test
Statistical Analysis 4: Comparison: ETOR 50 DMSO vs Placebo (Pt 2); Treatment comparison of Day 11 PGART frequencies (ETOR 50 DMSO vs Placebo [Pt 2]) was performed using a two-sided Jonckheere-Terpstra test; Test type: Superiority or Other; p = 0.3992, Jonckheere-Terpstra test
Statistical Analysis 5: Comparison: ETOR 50 DMSO vs Placebo (Pt 2); Treatment comparison of Day 14 PGART frequencies (ETOR 50 DMSO vs Placebo [Pt 2]) was performed using a two-sided Jonckheere-Terpstra test; Test type: Superiority or Other; p = 0.6626, Jonckheere-Terpstra test
Statistical Analysis 6: Comparison: ETOR 50 DMSO vs Placebo (Pt 2); Treatment comparison of post-trial PGART frequencies (ETOR 50 DMSO vs Placebo [Pt 2]) was performed using a two-sided Jonckheere-Terpstra test; Test type: Superiority or Other; p = 0.3150, Jonckheere-Terpstra test

8. Secondary Outcome: Study Parts 1 and 2: Number of Participants Who Experienced at Least One Adverse Event
Description: An adverse event is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure.
Time Frame: Study Part 1: up to Day 47; Study Part 2: up to Day 28
Population: Safety analysis set defined as all treated participants (etoricoxib or placebo) based on the treatment received rather than the randomized assignment.
Measure: Number; unit: Participants
Groups:
- ETOR 75 PG (Pt 1): Single-dose etoricoxib 75 mg (2.15 mL) 4% PG gel applied topically.
- ETOR 150 DMSO (Pt 1): Single-dose etoricoxib 150 mg (3.94 mL) 4% DMSO gel applied topically.
- ETOR 150 PG (Pt 1): Single-dose etoricoxib 150 mg (4.30 mL) 4% PG gel applied topically.
- ETOR OD (Pt 1): Single-dose etoricoxib 163 mg (4.30 mL) 4% DMSO gel applied topically (DMSO formulation administered in overdose/error).
- ETOR 50 DMSO (Pt 2): Etoricoxib 50 mg (1.31 mL, 4% DMSO gel) applied topically twice daily to the affected knee for a period of 2 weeks.
Arm/Group | ETOR 75 DMSO | ETOR 75 PG (Pt 1) | ETOR 150 DMSO (Pt 1) | ETOR 150 PG (Pt 1) | ETOR OD (Pt 1) | Placebo (Pt 1) (Deviation) | ETOR 50 DMSO (Pt 2) | Placebo (Pt 2)
Number analyzed (Participants) | 20 | 20 | 20 | 18 | 2 | 2 | 24 | 24
Participants | 1 | 1 | 1 | 1 | 2 | 0 | 6 | 5

9. Secondary Outcome: Study Parts 1 and 2: Number of Participants Who Discontinued Study Drug Due to an Adverse Event
Description: as for outcome 8
Time Frame: Study Part 1: up to Day 47; Study Part 2: up to Day 28
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | ETOR 75 DMSO | ETOR 75 PG (Pt 1) | ETOR 150 DMSO (Pt 1) | ETOR 150 PG (Pt 1) | ETOR OD (Pt 1) | Placebo (Pt 1) (Deviation) | ETOR 50 DMSO (Pt 2) | Placebo (Pt 2)
Number analyzed (Participants) | 20 | 20 | 20 | 18 | 2 | 2 | 24 | 24
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Study Part 1: up to Day 47; Study Part 2: up to Day 28
Description: An adverse event is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure.
Groups:
- ETOR 75 DMSO (Pt 1): Single-dose etoricoxib 75 mg (1.97 mL) 4% DMSO gel applied topically.
Arm/Group | ETOR 75 DMSO (Pt 1) | ETOR 75 PG (Pt 1) | ETOR 150 DMSO (Pt 1) | ETOR 150 PG (Pt 1) | ETOR OD (Pt 1) | Placebo (Pt 1) (Deviation) | ETOR 50 DMSO (Pt 2) | Placebo (Pt 2)
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/18 | 0/2 | 0/2 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 1/18 | 2/2 | 0/2 | 2/24 | 2/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ETOR 75 DMSO (Pt 1) (N=20) | ETOR 75 PG (Pt 1) (N=20) | ETOR 150 DMSO (Pt 1) (N=20) | ETOR 150 PG (Pt 1) (N=18) | ETOR OD (Pt 1) (N=2) | Placebo (Pt 1) (Deviation) (N=2) | ETOR 50 DMSO (Pt 2) (N=24) | Placebo (Pt 2) (N=24)
Cholecystocholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.